CLINICAL TRIAL: NCT02955186
Title: Fyn Kinase Inhibitors and Alcohol Drinking
Brief Title: Saracatinib and Alcohol Drinking
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Suchitra Krishnan-Sarin, Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1601017043; 2P50AA012870-16 (NIH)
Record Dates: First submitted 2016-11-01; First posted 2016-11-04 (Estimated); Results first posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Alcohol Drinking
MeSH Terms: conditions — Alcohol Drinking | interventions — saracatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 125 mg saracatinib (Experimental): Participants will take 125 mg of saracatinib daily for 8 days.
  Interventions: Drug: Saracatinib
- Placebo (Placebo Comparator): Participants will take placebo daily for 8 days.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Saracatinib — Saracatinib 125 mg once per day for 8 days
  Other Names: AZD0530
  Arms: 125 mg saracatinib
Drug: Placebos — Placebo once per day for 8 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effects of the study medication, saracatinib/AZD0530 (placebo or 125 mg/day) on alcohol drinking behavior in a laboratory setting in which participants are given an initial drink of alcohol followed by the choice to drink up to 12 more drinks over a three-hour period. The investigators hypothesize that saracatinib will reduce craving and number of drinks consumed prior to and after exposure to the initial drink of alcohol and during the three hour drinking period.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-50
* Able to read English at 6th grade level or higher and to complete study evaluations
* Regular alcohol drinker

Exclusion Criteria:

* Individuals who are seeking alcohol treatment
* Medical conditions that would contraindicate the use of saracatinib
* Regular use of other substances

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-09 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-06-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CMHC, Substance Abuse Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 54 participants agreed to the study but 4 did not end up participating in the full study and were never randomized to treatment.
Period: Overall Study
Arm/Group | 125 mg Saracatinib | Placebo
Started | 33 | 17
Completed | 26 | 15
Not Completed | 7 | 2
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 125 mg Saracatinib | Placebo | Total
Number analyzed (Participants) | 33 | 17 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (7.8) | 30 (7.9) | 29 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 25
  Male | 16 | 9 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 6 | 17
  White | 21 | 10 | 31
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 17 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Drinks Consumed From Baseline to Day 8 (Minus Baseline)
Description: Change in the number of standard drinks consumed at the drinking session (ADP 2) after taking study medication minus the number of standard drinks consumed at baseline (ADP 1).
Time Frame: Baseline and Day 8
Measure: Least Squares Mean (Standard Error); unit: drinks
Arm/Group | 125 mg Saracatinib | Placebo
Number analyzed (Participants) | 26 | 15
drinks | -1.85 (.75) | -2.33 (.99)

2. Primary Outcome: Craving-Baseline Adjusted Total Area Under the Curve (AUC) During the Drinking Session Using the YCS
Description: Craving for alcohol based on Yale Craving Scale (YCS), scores ranging from 0-112 mm on a visual analog scale, with higher measurements indicating higher craving. The baseline-adjusted craving is change score from baseline at Day 7.
Time Frame: Baseline and Day 7
Measure: Least Squares Mean (Standard Error); unit: units on a scale*days
Arm/Group | 125 mg Saracatinib | Placebo
Number analyzed (Participants) | 33 | 17
units on a scale*days | 3133 (371) | 2876 (489)

3. Secondary Outcome: Area Under the Curve (AUC) During the Drinking Session Using the Stimulation Responses to Alcohol (BAES)
Description: Biphasic Alcohol Effects Scale (BAES) scores will be used to assess stimulation. The scale ranges from 0-70, with a higher score indicating more sedated.
Time Frame: Day 8 Adlib
Measure: Mean (Standard Deviation); unit: units on a scale*days
Arm/Group | 125 mg Saracatinib | Placebo
Number analyzed (Participants) | 33 | 17
units on a scale*days | 1650.8 (2185.7) | 1607.1 (1984.3)

4. Secondary Outcome: Area Under the Curve (AUC) During the Drinking Session Using the Sedation Responses to Alcohol (BAES)
Description: Biphasic Alcohol Effects Scale (BAES) scores will be used to assess sedation. The scale ranges from 0-70, with a higher score indicating more sedated.
Time Frame: Day 8 Adlib
Measure: Mean (Standard Deviation); unit: units on a scale*days
Arm/Group | 125 mg Saracatinib | Placebo
Number analyzed (Participants) | 33 | 17
units on a scale*days | 1149.9 (1495.5) | 515.29 (551)

ADVERSE EVENTS:
Time Frame: Adverse Event data were collected at baseline, daily during the 8 days of medication and then at one month follow-up.
Description: Adverse events were collected multiple times throughout the study: at baseline, daily during medication dosing, and one month following completion of study.
Arm/Group | 125 mg Saracatinib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/17
Other Adverse Events (participants affected / at risk) | 21/33 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 125 mg Saracatinib (N=33) | Placebo (N=17)
car accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 125 mg Saracatinib (N=33) | Placebo (N=17)
Abdominal Pain (Gastrointestinal disorders) | 3 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 5 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Fatigue (Psychiatric disorders) | 2 | 3
Headache (Nervous system disorders) | 5 | 1
Cold symptoms (Ear and labyrinth disorders) | 6 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Joint Pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 2 | 2
Sore throat (Ear and labyrinth disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
High feeling (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/86/NCT02955186/Prot_SAP_000.pdf